CLINICAL TRIAL: NCT04192591
Title: A 5-year Superion™ IDS Clinical Outcomes Post-Approval Evaluation (SCOPE)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4082
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Lumbar Spinal Stenosis; LSS; Chronic Pain; Leg Pain
MeSH Terms: conditions — Spinal Stenosis; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Superion™ IDS device (Experimental): Superion™ Indirect Decompression System (IDS)
  Interventions: Device: Superion™ IDS device

INTERVENTIONS:
Device: Superion™ IDS device — The Superion™ IDS is a minimally-invasive spinal implant that treats LSS symptoms by limiting extension at the symptomatic level that compresses the neural elements and is designed for percutaneous surgical placement.

SUMMARY:
To compile real-world outcomes of the Superion™ IDS in routine clinical practice.

DETAILED DESCRIPTION:
To compile real-world outcomes of the Superion™ IDS in routine clinical practice, when used according to the applicable Directions for Use

ELIGIBILITY:
Key Inclusion Criteria:

* 45 years of age or older when written informed consent is obtained
* Persistent leg/buttock/groin pain, with or without back pain that is consistently relieved by flexion activities (example: sitting or bending over a shopping cart).
* Diagnosis of degenerative spinal stenosis of the lumbar spine, defined as the narrowing of the midline sagittal spinal canal (central) and/or narrowing between the facet superior articulating process (SAP), the posterior vertebral margin (lateral access), and the nerve root canal (foraminal).
* Subject signed a valid, IRB-approved informed consent form (ICF) provided in English.
* Subjects, who, in the opinion of the Clinical Investigator, are able to understand this clinical investigation, cooperate with the investigational procedures and are willing to return for all the required post-treatment follow-ups.
* Able to independently read and complete all questionnaires and assessments provided in English

Key Exclusion Criteria:

* Axial back pain only.
* Fixed motor deficit in lower extremity(ies) due to LSS.
* Has any pain-related diagnosis, medical/psychological condition or external factors that, in the investigator's medical judgment, might confound reporting of study outcomes (e.g. history of pelvic pain, anginal pain, chronic migraine, involved in litigation, workmen's compensation, spinal tumor)
* Participating (or intends to participate) in another drug or device clinical trial that may influence the data that will be collected for this study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2038-02 (Estimated); Study Completion 2041-02 (Estimated)

PRIMARY OUTCOMES:
Rate of success at the 24-month follow-up visit | 24-Months
  Non-inferiority of overall subject success at the 24-Month visit vs. the 24-month visit in IDE trial. An individual subject will be considered a success if they meet all of the following conditions at the 24-month follow-up visit:
  1. Clinically significant improvement of neurogenic claudication symptoms as determined by meeting at least two of three domains of the ZCQ
     * ≥ 0.5-point improvement in physical function
     * ≥ 0.5-point improvement in symptom severity
     * ≤ 2.5 point on patient satisfaction domain
  2. No reoperations, removals, revisions, or supplemental fixation at the index level(s)
  3. No major implant or procedure-related complications
     * no dislodgement, migration, or device deformation
     * no new or persistent worsened neurological deficit at the index level†
     * no unhealed spinous process fractures † Defined as a serious adverse event wherein there is any new/worsening of motor or sensory function at 12 months, compared to baseline, which persists to 24 months

SECONDARY OUTCOMES:
Patient Satisfaction: VertiFlex® Patient Satisfaction Survey | 24-, 36-, 48- and 60-Months
  Proportion of subjects with VertiFlex® Patient Satisfaction Survey scoring ≥3 on a 4-point scale

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Bloom Lyons, Study Director — Boston Scientific Corporation
Locations (23):
- United States (23):
  - Coastal Research Institute, LLC, Carlsbad, California
  - MarinHealth Spine Institute, Larkspur, California
  - Vitamed Research, Rancho Mirage, California
  - IPM Medical Group Inc., Walnut Creek, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - The Orthopaedic Institute, Gainesville, Florida
  - Alliance Spine and Pain Centers, Atlanta, Georgia
  - Centurion Spine and Pain, Waycross, Georgia
  - North Idaho Day Surgery, Post Falls, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Ascension Alexian Brothers, Elk Grove Village, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - Neuroscience Research Center, LLC, Overland Park, Kansas
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Michigan Pain Specialists, Ypsilanti, Michigan
  - Weill Cornell Medical University, New York, New York
  - Pacific Sports and Spine, LLC, Eugene, Oregon
  - Center for Interventional Pain and Spine, Lancaster, Pennsylvania
  - SC Pain and Spine Specialists, Murrells Inlet, South Carolina
  - Precision Spine Care, Tyler, Texas
  - Swedish Health Services, Seattle, Washington
  - Northwest Pain Care, Spokane, Washington
  - The Spine and Nerve Center of Saint Francis Hospital, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No